CLINICAL TRIAL: NCT04474691
Title: staRt: Enhancing Speech Treatment With Smartphone-delivered Biofeedback
Acronym: staRt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: staRt single-case; R41DC016778 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-07-17 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2021-12

CONDITIONS: Speech Sound Disorder
Keywords: speech; articulation; motor development
MeSH Terms: conditions — Speech Sound Disorder; Speech

STUDY DESIGN:
Intervention Model Description: Children with /r/ misarticulation will receive 16 sessions/8 weeks of intervention using staRt. Individual sessions will be randomly assigned to include the visual biofeedback display (visual-acoustic biofeedback treatment) or exclude it (traditional treatment). Participants will receive an equal number of sessions (8) of each type.
Who Masked: Outcomes Assessor
Masking Description: Acoustic measures will be obtained by research assistants blinded to the treatment condition assigned for each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual-acoustic biofeedback (Experimental)
  Interventions: Behavioral: Visual-acoustic biofeedback
- Traditional articulation treatment (Active Comparator)
  Interventions: Behavioral: Traditional articulation treatment

INTERVENTIONS:
Behavioral: Traditional articulation treatment — Traditional articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract can be used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available. Knowledge of performance feedback could describe either the desired articulator placement or the auditory quality of the target sound.
  Arms: Traditional articulation treatment
Behavioral: Visual-acoustic biofeedback — In visual-acoustic biofeedback treatment, the elements of traditional treatment (auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum generated by the staRt app. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3. Knowledge of performance feedback will typically involve reference to the location of the third peak or 'bump' on the visual display.
  Arms: Visual-acoustic biofeedback

SUMMARY:
Previous research suggests that biofeedback can outperform traditional interventions for RSE, but no controlled studies have tested this hypothesis in the context of app-delivered biofeedback. The objective of this aim is to use the staRt app to test our working hypothesis that speakers will make larger gains in /r/ accuracy when app-based treatment incorporates biofeedback, compared to a non-biofeedback condition. With a network of cooperating SLPs, this project will recruit 15 children with /r/ misarticulation to receive 8 weeks of intervention using staRt. Individual sessions will be randomly assigned to include or exclude the visual biofeedback display. Randomization tests will be used to evaluate, for each individual, whether larger increments of change are associated with biofeedback and non-biofeedback sessions.

ELIGIBILITY:
Inclusion Criteria:

* Normal performance on a pure-tone hearing screening at 20 dB HL, a screening examination of oral-motor structure and function, and a test of receptive language.

Exclusion Criteria:

* History of major behavioral, neurological, or hearing impairment, per parent and/or SLP report.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Social media and mailing lists were used to identify certified speech-language pathologists interested in providing the study treatment to consenting participants on their caseload. Clinical partners completed CITI human subjects training (both basic social/behavioral and Good Clinical Practice). They were also required to complete an Individual Investigator Agreement (if not already covered by an existing IRB) or secure a reliance agreement (if covered by an existing IRB) with the IRB at NYU.
Pre-assignment Details: This study used a within-subjects design. Each participant received both treatment conditions, with sessions randomly assigned to feature one condition or the other.
Units Other Than Participants: Sessions
Groups:
- Visual-acoustic Biofeedback and Traditional Articulation Treatment: Visual-acoustic biofeedback: In visual-acoustic biofeedback treatment, the elements of traditional treatment (auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum generated by the staRt app. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3. Knowledge of performance feedback will typically involve reference to the location of the third peak or 'bump' on the visual display.
  Traditional articulation treatment: Traditional articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract can be used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available. Knowledge of performance feedback could describe either the desired articulator placement or the auditory quality of the target sound.
Period: Overall Study
Arm/Group | Visual-acoustic Biofeedback and Traditional Articulation Treatment
Started | 15; 240 Sessions (The number reported refers to the number of sessions scheduled across all participants.)
Visual-acoustic Biofeedback | 8; 56 Sessions (The number reported refers to the number of sessions completed across all participants.)
Traditional Articulation Treatment | 8; 53 Sessions (The number reported refers to the number of sessions completed across all participants.)
Completed | 6; 96 Sessions (The number reported refers to the number of sessions completed across all participants.)
Not Completed | 9; 144 Sessions
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Groups:
- Visual-acoustic Biofeedback and Traditional Articulation Treatment: This study used a within-subjects design. Each participant received two treatment conditions (visual-acoustic biofeedback and ultrasound biofeedback), with sessions randomly assigned to feature one condition or the other. In traditional articulation treatment, the clinician provides auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract can be used as visual aids; however, no real-time visual display of articulatory or acoustic information is made available. Knowledge of performance feedback could describe either the desired articulator placement or the auditory quality of the target sound. In visual-acoustic biofeedback treatment, the elements of traditional articulatory treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants are cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency.
Arm/Group | Visual-acoustic Biofeedback and Traditional Articulation Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: F3-F2 Distance, an Acoustic Measure That Correlates With Perceptual Accuracy of /r/, Measured From /r/ Sounds Produced in Treatment Sessions.
Description: From recordings of words containing /r/ produced during treatment sessions, the sound /r/ was flagged for measurement and the first three formants (F1, F2, F3) were extracted from the center of the /r/ interval. The distance between the second and third formants (F3-F2) was used as the index of rhoticity. F3-F2 is small in perceptually accurate /r/, larger values indicate lower accuracy. Summary statistics report the mean and standard deviation of normalized F3-F2 distance for each treatment condition, pooled across participants and sessions. A two-tailed paired-samples t-test (superiority criterion) was used to compare mean F3-F2 distance for each treatment condition across subjects.
Time Frame: F3-F2 distance was measured in all 16 treatment sessions (eight of each type), which were administered over eight weeks.
Population: Note that this study used a within-subjects design. Each participant received both treatment conditions, with individual sessions randomly assigned to feature one condition or the other.
Measure: Mean (Standard Deviation); unit: Hz
Groups:
- Traditional Articulation Treatment: In traditional articulation treatment, the clinician provides auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract can be used as visual aids; however, no real-time visual display of articulatory or acoustic information is made available. Knowledge of performance feedback could describe either the desired articulator placement or the auditory quality of the target sound.
- Visual-acoustic Biofeedback: In visual-acoustic biofeedback treatment, the elements of traditional articulatory treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants are cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency.
Arm/Group | Traditional Articulation Treatment | Visual-acoustic Biofeedback
Number analyzed (Participants) | 6 | 6
Hz | 1793.3 (158.3) | 1772.2 (99.5)
Statistical Analysis 1: Comparison: Traditional Articulation Treatment; Test type: Superiority; p = .67, t-test, 1 sided; df = 7; Mean Difference (Final Values) = 21.1 — Traditional treatment condition - visual-acoustic biofeedback treatment condition. Because more accurate productions have lower acoustic values, a positive difference would indicate an advantage for biofeedback

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The definition of adverse event and serious adverse event used to collect adverse event information does not differ from that of clinicaltrials.gov.
Arm/Group | Visual-acoustic Biofeedback | Traditional Articulation Treatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04474691/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04474691/SAP_001.pdf